CLINICAL TRIAL: NCT04180787
Title: Effects of a Caffeine- and Protein-Containing Coffee Beverage on Metabolism and Muscular Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: Vital Pharmaceuticals, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 20-0130
Record Dates: First submitted 2019-11-20; First posted 2019-11-29 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Exercise Performance; Metabolism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Keto Coffee (Experimental): VPX Bang® Keto Coffee beverage
  Interventions: Dietary Supplement: Beverage Consumption
- Placebo (Placebo Comparator): Flavor-matched placebo beverage
  Interventions: Dietary Supplement: Beverage Consumption

INTERVENTIONS:
Dietary Supplement: Beverage Consumption — Participants will consume either VPX Bang® Keto Coffee beverage or flavor-matched placebo beverage in each condition.

SUMMARY:
The purpose of this randomized, double-blind, crossover study is to investigate the effects of Bang® Keto Coffee on resting and post-exercise metabolism and muscular performance during lower body resistance exercise.

DETAILED DESCRIPTION:
Resistance-trained males and females will be recruited for participation in a randomized, double-bind, crossover trial. After providing informed consent, each participant will undergo a familiarization session to become accustomed to the study procedures. Following familiarization, each participant will complete two laboratory visits consisting of metabolism and exercise performance assessments. In both visits, a baseline assessment of resting metabolic rate (RMR) and respiratory exchange ratio (RER) will be conducted using indirect calorimetry. Following the initial RMR assessment, each participant will ingest a coffee flavored beverage, either VPX Bang® Keto Coffee or a flavor-matched placebo. After beverage consumption, the participant will return to the supine position and rest prior to initiation of the second RMR assessment. Immediately following the second RMR assessment, the participant will begin a 5-minute dynamic bodyweight warm up. Participants will then begin squat testing procedures on a mechanized squat device. After completing the squat testing, participants will complete a standard 1-repetition maximum and repetitions to failure using a plate-loaded hip sled machine. Following the hip sled testing, participants will repeat the mechanized squat testing. Following completion of the exercise testing, a third and final RMR assessment will be performed. Following successful completion of the first condition, each participant will enter a wash out period, after which the visit will be repeated with ingestion of the alternative beverage.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 40
* Generally healthy (defined as an absence of any disease or medical condition which could potentially be negatively affected by consumption of the commercially available dietary supplement of performance of exercise, including but not limited to musculoskeletal or cardiovascular diseases).
* Resistance-trained, defined as completing 3+ resistance training sessions per week for at least one year and including at least weekly training of the lower body through a multi-joint exercise such as the squat or leg press.
* Regular caffeine consumption, defined as an average self-reported daily intake of 200+ mg of caffeine, which is equivalent to approximately 2 cups of coffee.

Exclusion Criteria:

* Failing to meet any of the aforementioned inclusion criteria.
* Pregnant or breastfeeding (for female participants)
* Taking prescription medication which could reasonably make participation unsafe for the participant or influence study outcomes
* An inability to complete lower body resistance exercise due to injury or medical condition
* Self-reported caffeine sensitivity, as indicated by unwanted side effects when caffeine is consumed.
* Allergy to any of the ingredients in the commercially available dietary supplement
* Self-reported claustrophobia (due to metabolism testing)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Isometric Force Production | Assessed approximately 45 minutes after beverage ingestion
  Isometric force production on mechanized squat device
Isometric Force Production | Assessed approximately 80 minutes after beverage ingestion
  Isometric force production on mechanized squat device
Isokinetic Force Production | Assessed approximately 45 minutes after beverage ingestion
  Isokinetic force production on mechanized squat device
Isokinetic Force Production | Assessed approximately 80 minutes after beverage ingestion
  Isokinetic force production on mechanized squat device.
Maximal Lower Body Strength | Assessed approximately 75 minutes after beverage ingestion
  One-repetition maximum on hip sled machine
Maximal Lower Body Endurance | Assessed approximately 75 minutes after beverage ingestion (following maximal lower body strength testing)
  Repetitions to failure on hip sled machine
Change in Metabolic Rate | Change in metabolic rate between: 1) before beverage ingestion (baseline) and 2) beginning approximately 10 minutes after completion of beverage ingestion
  Metabolic rate assessed via indirect calorimetry
Change in Metabolic Rate | Change in metabolic rate between: 1) before beverage ingestion (baseline) and 2) beginning approximately 5 minutes after completion of all exercise testing
  Metabolic rate assessed via indirect calorimetry
Change in Respiratory Exchange Ratio | Change in respiratory exchange ratio between: 1) before beverage ingestion (baseline) and 2) beginning approximately 10 minutes after completion of beverage ingestion
  Respiratory exchange ratio as assessed via indirect calorimetry
Change in Respiratory Exchange Ratio | Change in respiratory exchange ratio between: 1) before beverage ingestion (baseline) and 2) beginning approximately 5 minutes after completion of all exercise testing.
  Respiratory exchange ratio as assessed via indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Grant M Tinsley, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Department of Kinesiology & Sport Management, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Harty PS, Stratton MT, Escalante G, Rodriguez C, Dellinger JR, Williams AD, White SJ, Smith RW, Johnson BA, Sanders MB, Tinsley GM. Effects of Bang(R) Keto Coffee Energy Drink on Metabolism and Exercise Performance in Resistance-Trained Adults: A Randomized, Double-blind, Placebo-controlled, Crossover Study. J Int Soc Sports Nutr. 2020 Aug 24;17(1):45. doi: 10.1186/s12970-020-00374-5. PMID 32831109